CLINICAL TRIAL: NCT05152758
Title: STABILITY: Physical Activity Intervention at 7 Years Post-Anterior Cruciate Ligament Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STABILITY PARx Sub-Study
Record Dates: First submitted 2021-11-04; First posted 2021-12-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Post-traumatic Osteoarthritis
Keywords: physical activity; anterior cruciate ligament reconstruction; osteoarthritis
MeSH Terms: conditions — Motor Activity; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This trial will randomize up to 196 ACL-reconstruction patients to receive either the standard of care or a physical activity prescription (PARx) at 7 years post-reconstruction in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patients will receive the usual care.
- Physical Activity Prescription (PARx) (Experimental): Patients will be prescribed technology-based physical activity programming.
  Interventions: Device: PARx

INTERVENTIONS:
Device: PARx — Prescription Physical Activity Programming Application
  Arms: Physical Activity Prescription (PARx)

SUMMARY:
Anterior cruciate ligament (ACL) ruptures are very common knee injuries amongst youth involved in sports and are often treated through ACL reconstruction surgeries. Unfortunately, up to 50% of individuals who undergo ACL reconstruction develop post-traumatic osteoarthritis (PTOA) in their injured knee by 20 years post-reconstruction causing pain, decreasing mobility, and impacting quality of life in young active individuals. Much remains unknown regarding the secondary prevention of PTOA, and more investigation is necessary to better understand its disease progression post-ACL reconstruction and types of conservative interventions that can prevent or delay its onset.

Physical activity has improved patient-reported outcomes across many different chronic diseases including knee osteoarthritis (OA), and physical activity prescription has been shown to be an effective way to increase patients' levels of physical activity. It has not yet been heavily investigated in the context of post-ACL reconstruction, and individuals often exhibit decreased physical activity after ACL reconstruction which causes suboptimal cartilage health. Thus, physical activity prescription may improve habitual joint loading, leading to improved cartilage health and patient-reported health outcomes.

DETAILED DESCRIPTION:
ACL injuries are extremely common knee injuries sustained by athletes participating in sports involving sudden changes of direction like jumping, cutting and pivoting. Every year, approximately 1 in 3500 individuals injure their ACL. ACL reconstruction surgery is a popular treatment option for young athletes that aims to re-establish knee stability and restore function, enabling high rates of return to sport. Unfortunately, despite reconstruction surgery's short-term benefits, it does not significantly alter the course of post-traumatic osteoarthritis (PTOA) that often develops after sustaining a severe knee injury. In fact, over half of ACL patients present radiographic signs of OA by 20 years post-reconstruction surgery. Individuals with OA often have significantly impaired mobility, functionality, and quality of life, so appropriate rehabilitation protocols and conservative joint management strategies are necessary to improve knee health outcomes post-reconstruction and keep these patients healthy and active for as long as possible.

Physical activity has widely known preventive and therapeutic effects across many chronic diseases such as diabetes, hypertension, heart disease, and obesity. Similarly, there is widespread evidence of high physical activity levels reducing pain and increasing function and health-related quality of life in individuals with knee and hip osteoarthritis, indicating its efficacy as a conservative measure for improving joint health. In contrast, sedentary behaviour increases the risk of OA development and other comorbidities by increasing body mass index (BMI), causing poorer cartilage health, reducing muscle quality, and increasing systemic inflammation. Following ACL reconstruction, individuals are susceptible to adopting more sedentary lifestyles due to a fear of re-injury through movement, evidenced by relatively lower self-reported physical activity levels compared to before injury. While ACL injuries may initiate OA pathogenesis, sedentary behaviour is a modifiable risk factor that can further facilitate disease progression. Since physical activity prescription effectively increases physical activity levels, it offers potential utility for improving knee joint health post-reconstruction surgery and preventing or delaying the onset of PTOA.

Objectives:

1. To examine the effects of physical activity prescription on patient-reported outcomes (KOOS and IKDC scores)
2. To examine the effects of physical activity prescription on femoral trochlear cartilage thickness and echo intensity based on ultrasound imaging over 1 year.
3. To analyze the impact of patients' gait biomechanics on changes in patient-reported outcomes and femoral trochlear cartilage health outcomes due to the physical activity intervention.

Hypotheses:

1. Those assigned to the physical activity prescription group will have higher KOOS and IKDC scores than those in the control group following 1 year.
2. Physical activity prescription will lead to less reductions in echo intensity and heterogeneity of the femoral trochlear cartilage over 1 year.
3. Poorer femoral trochlear cartilage health imaging outcomes (greater reductions in echo intensity and heterogeneity) and lower KOOS and IKDC scores at 1 year will be associated with larger vertical ground reaction forces, smaller knee flexion angles, greater knee adduction moments, smaller knee extensor moments, and larger vertical loading rates of the involved limb.

ELIGIBILITY:
Inclusion Criteria:

* Subjects following up for 7-year visits as part of the Standard ACL Reconstruction vs ACL + Lateral Extra-Articular Tenodesis Study (STAbiLiTY)

Exclusion Criteria:

* Unable/unwilling to follow up for the study period
* Does not have access to the internet and/or smartphone
* Cannot communicate in English
* Unstable medical conditions that would preclude engagement in prescribed physical activity
* Scheduled for second surgery over study period

Ages: 21 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) | Baseline
  This form uses a subjective scale to provide a score from 0 to 100 indicating the patient's overall level of function. The total score is determined by adding individual scores from three categories: symptoms, sports activity, and knee function.
International Knee Documentation Committee (IKDC) | 2 months
  This form uses a subjective scale to provide a score from 0 to 100 indicating the patient's overall level of function. The total score is determined by adding individual scores from three categories: symptoms, sports activity, and knee function.
International Knee Documentation Committee (IKDC) | 6 months
  This form uses a subjective scale to provide a score from 0 to 100 indicating the patient's overall level of function. The total score is determined by adding individual scores from three categories: symptoms, sports activity, and knee function.
International Knee Documentation Committee (IKDC) | 12 months
  This form uses a subjective scale to provide a score from 0 to 100 indicating the patient's overall level of function. The total score is determined by adding individual scores from three categories: symptoms, sports activity, and knee function.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee Injury and Osteoarthritis Outcome Score | 2 months
  Knee-specific survey that evaluates short-term and long-term consequences of knee injury with 42 questions across 5 subscales: pain, other symptoms, function in daily living, function in sport and recreation, and knee-related quality of life. Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee Injury and Osteoarthritis Outcome Score | 6 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee Injury and Osteoarthritis Outcome Score | 12 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Ultrasonographic Femoral Trochlear Cartilage Imaging | Baseline
  Ultrasonographic imaging of the femoral trochlear cartilage will help visualize and compare deleterious cartilage changes between the PA intervention group and the usual care group. A Logiq e ultrasound machine (GE Healthcare) will be used to measure cartilage thickness, echo-intensity, and heterogeneity to assess composition quality.
Ultrasonographic Femoral Trochlear Cartilage Imaging | 12 months
  Ultrasonographic imaging of the femoral trochlear cartilage will help visualize and compare deleterious cartilage changes between the PA intervention group and the usual care group. A Logiq e ultrasound machine (GE Healthcare) will be used to measure cartilage thickness, echo-intensity, and heterogeneity to assess composition quality.
Physical Activity Evaluation using Global Physical Activity Questionnaire (GPAQ) and MyRecovery app | Baseline
  The GPAQ is a 22-item questionnaire designed to estimate patients' physical activity levels in work, transport, and leisure time as well as time spent doing sedentary behaviours. It also asks two questions to determine the patient's level of positive attitude towards physical activity and the barriers that may prevent them from physical activity engagement. MyRecovery is a smartphone app that tracks steps per day, light/moderate/vigorous activity, and total MET-min through accelerometer data.
Physical Activity Evaluation using Global Physical Activity Questionnaire (GPAQ) and MyRecovery app | 2 months
  The GPAQ is a 22-item questionnaire designed to estimate patients' physical activity levels in work, transport, and leisure time as well as time spent doing sedentary behaviours. It also asks two questions to determine the patient's level of positive attitude towards physical activity and the barriers that may prevent them from physical activity engagement. MyRecovery is a smartphone app that tracks steps per day, light/moderate/vigorous activity, and total metabolic equivalents through accelerometer data.
Physical Activity Evaluation using Global Physical Activity Questionnaire (GPAQ) and MyRecovery app | 6 months
  The GPAQ is a 22-item questionnaire designed to estimate patients' physical activity levels in work, transport, and leisure time as well as time spent doing sedentary behaviours. It also asks two questions to determine the patient's level of positive attitude towards physical activity and the barriers that may prevent them from physical activity engagement. MyRecovery is a smartphone app that tracks steps per day, light/moderate/vigorous activity, and total metabolic equivalents through accelerometer data.
Physical Activity Evaluation using Global Physical Activity Questionnaire (GPAQ) and MyRecovery app | 12 months
  The GPAQ is a 22-item questionnaire designed to estimate patients' physical activity levels in work, transport, and leisure time as well as time spent doing sedentary behaviours. It also asks two questions to determine the patient's level of positive attitude towards physical activity and the barriers that may prevent them from physical activity engagement. MyRecovery is a smartphone app that tracks steps per day, light/moderate/vigorous activity, and total MET-min through accelerometer data.
Three-dimensional Motion-captured Gait Biomechanics Analysis | Baseline
  Walking gait biomechanics will be motion-captured and analyzed to identify individuals with asymmetries in lower-limb biomechanics during walking. Metrics used will include peak knee adduction moment, peak knee flexion moment, vertical ground reaction force, and vertical loading rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Thornton, MD PhD, Principal Investigator — Western University
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cinque ME, Dornan GJ, Chahla J, Moatshe G, LaPrade RF. High Rates of Osteoarthritis Develop After Anterior Cruciate Ligament Surgery: An Analysis of 4108 Patients. Am J Sports Med. 2018 Jul;46(8):2011-2019. doi: 10.1177/0363546517730072. Epub 2017 Oct 6. PMID 28982255
- [Background] Ravalli S, Castrogiovanni P, Musumeci G. Exercise as medicine to be prescribed in osteoarthritis. World J Orthop. 2019 Jul 18;10(7):262-267. doi: 10.5312/wjo.v10.i7.262. eCollection 2019 Jul 18. PMID 31363456
- [Background] Evans J, Nielson JL. Anterior Cruciate Ligament Knee Injuries. 2021 Feb 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2021 Jan-. PMID: 29763023.
- [Background] Kraus VB, Sprow K, Powell KE, Buchner D, Bloodgood B, Piercy K, George SM, Kraus WE; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Effects of Physical Activity in Knee and Hip Osteoarthritis: A Systematic Umbrella Review. Med Sci Sports Exerc. 2019 Jun;51(6):1324-1339. doi: 10.1249/MSS.0000000000001944. PMID 31095089
- [Background] Maly MR, Marriott KA, Chopp-Hurley JN. Osteoarthritis year in review 2019: rehabilitation and outcomes. Osteoarthritis Cartilage. 2020 Mar;28(3):249-266. doi: 10.1016/j.joca.2019.11.008. Epub 2019 Dec 23. PMID 31877379
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383